CLINICAL TRIAL: NCT01422395
Title: A Study to Compare Vitrified/Warmed Oocytes vs. Fresh Sibling Oocytes Collected Following Controlled Ovarian Stimulation Using Follistim AQ and Ganirelix Acetate on Fertilization Rates, Zygote Quality, Embryo Quality and Embryo Development
Brief Title: Effect of Oocyte Vitrification on Fertilization Rate, Embryo Quality and Development
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Main Line Fertility Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: MLFC-001
Record Dates: First submitted 2011-08-22; First posted 2011-08-24 (Estimated); Last update posted 2014-06-04 (Estimated); Status verified 2014-06

CONDITIONS: Fertility
Keywords: Vitrification; Egg Freezing; Oocyte Cryopreservation
MeSH Terms: interventions — Freezing

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- freezing (Experimental)
  Interventions: Procedure: Freezing
- No freezing (No Intervention)

INTERVENTIONS:
Procedure: Freezing — Vitrification
  Arms: freezing

SUMMARY:
Indications for oocyte (egg) vitrification (fast freezing) include the preservation of reproductive competence of young cancer patients who need chemotherapy, pelvic radiation, or surgical removal of ovaries for treatment. Furthermore, the ability to freeze oocytes allows patients to reduce the number of embryos frozen, thereby circumventing the moral and ethical dilemmas of having left-over embryos in cryostorage. In addition, oocyte cryopreservation could allow women to delay childbearing if they want or need to. Until recently, conventional cryopreservation protocols have remained too inefficient for practical application in an infertility center. Very little is known about the effects of vitrification on oocytes and subsequent embryo development, especially using the sibling model (group of oocytes from the same cohort of ovarian follicles within patient). The purpose of this study is to examine the effect of oocyte vitrification on fertilization rates, embryo quality and development.

ELIGIBILITY:
Inclusion Criteria:

* healthy women ages 21-37 (inclusive)undergoing IVF in an attempt to achieve pregnancy
* Day 2-4 FSH < 10 IU/ml, LH <12 IU/ml, and E2 <50 pg/ml
* Antimullerian Hormone (AMH) >1.5
* Between 5 and 20 basal antral follicles on day 2-4 of the menstrual cycle
* BMI >18 and <32

Exclusion Criteria:

* Smokers
* Polycystic Ovarian Syndrome (PCO)

Ages: 21 Years to 37 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2011-08; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
fertilization rate | 18 hours after insemination
Embryo Quality | day 3 and day 5
Embryo Development | Day 3 and day 5

CONTACTS AND LOCATIONS:
Overall Officials: Glassner J Michael, M.D., Principal Investigator — Main Line Fertility Center; Sharon H. Anderson, Ph.D, Study Director — Main Line Fertility Center
Locations (1):
- Main Line Fertility Center, Bryn Mawr, Pennsylvania, United States